CLINICAL TRIAL: NCT05952206
Title: Ischemic and Bleeding Outcomes After Angiolite Stent Implantation and an Abbreviated Dual Antiplatelet Therapy. A 2x2 Factorial, All-comer, Multicenter, Randomized Controlled Trial: ANGIODAPT
Brief Title: Ischemic and Bleeding Outcomes After Angiolite Stent Implantation and an Abbreviated Dual Antiplatelet Therapy
Acronym: ANGIODAPT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ANGIODAPT-01
Record Dates: First submitted 2023-05-24; First posted 2023-07-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: angiolite; dual antiplatelet therapy; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, randomized (1:1:1:1), factorial design 2x2, active control, and multicentre clinical trial.
Masking Description: Masking:
  * Open-label for the stent type
  * Open-label for the antiplatelet regimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Angiolite and abbreviated DAPT (Experimental): Acute coronary syndrome patients:
  * Need for OAC: TAT + OAC for one week. Double therapy composed of clopidogrel + OAC up to 6 months.
  * No need for OAC: DAPT with acetylsalicylic acid + prasugrel or ticagrelor for 1M. Only the same P2Y12 inhibitor up to 12M.
  Chronic coronary syndrome patients:
  * Need for OAC: TAT + clopidogrel + OAC for one week. Double therapy composed of clopidogrel + OAC up to 6M.
  * No need for OAC: DAPT with acetylsalicylic acid + clopidogrel for one month. Only clopidogrel up to 12M.
  Interventions: Device: Angiolite: Sirolimus-eluting stent; Drug: 1-month DAPT
- Xience stent family and abbreviated DAPT (Experimental): Acute coronary syndrome patients:
  * Need for OAC: TAT + OAC for one week. Double therapy composed of clopidogrel + OAC up to 6M.
  * No need for OAC: DAPT with acetylsalicylic acid + prasugrel or ticagrelor for 1 month. Only the same P2Y12 inhibitor up to 12M.
  Chronic coronary syndrome patients:
  * Need for OAC: TAT + clopidogrel + OAC for one week. Double therapy composed of clopidogrel + OAC up to 6M.
  * No need for OAC: DAPT with acetylsalicylic acid + clopidogrel for one month. Only clopidogrel up to 12M.
  Interventions: Device: Xience: Everolimus-eluting stent; Drug: 1-month DAPT
- Angiolite and standard of care DAPT (Active Comparator): Acute coronary syndrome patients:
  * Need for OAC: Recommendations of the current ESC guideline: 1M of TAT (acetylsalicylic acid + clopidogrel + OAC). Dual therapy (acetylsalicylic acid or clopidogrel + OAC) up to 12M. If ischemic concerns prevail, TAT can be extended up to 6M and dual therapy up to 12M.
  * No need for OAC: Recommendations of the current ESC guideline: DAPT with acetylsalicylic acid and prasugrel or ticagrelor is recommended up to 12M.
  Chronic coronary syndrome:
  * Need for OAC: Recommendations of the current ESC guidelines: 1M of TAT (acetylsalicylic acid + clopidogrel + OAC). Dual therapy (acetylsalicylic acid or clopidogrel + OAC) up to 12M. If ischemic concerns prevail, TAT can be extended up to 6M and dual therapy up to 12M.
  * No need for OAC: Recommendations of the current ESC guidelines: DAPT composed of acetylsalicylic acid + clopidogrel up to 6M. Then, continue with acetylsalicylic acid.
  Interventions: Device: Angiolite: Sirolimus-eluting stent; Drug: 12-month DAPT (Standard of care)
- Xience stent family and standard of care DAPT (Active Comparator): Acute coronary syndrome patients:
  * Need for OAC: Recommendations of the current ESC guideline: 1M of TAT (acetylsalicylic acid + clopidogrel + OAC). Dual therapy (acetylsalicylic acid or clopidogrel + OAC) up to 12M. If ischemic concerns prevail, TAT can be extended up to 6M and dual therapy up to 12M.
  * No need for OAC: Recommendations of the current ESC guideline: DAPT with acetylsalicylic acid and prasugrel or ticagrelor is recommended up to 12M.
  Chronic coronary syndrome:
  * Need for OAC: Recommendations of the current ESC guidelines: 1M of TAT (acetylsalicylic acid + clopidogrel + OAC). Dual therapy (acetylsalicylic acid or clopidogrel + OAC) up to 12M. If ischemic concerns prevail, TAT can be extended up to 6M and dual therapy up to 12M.
  * No need for OAC: Recommendations of the current ESC guidelines: DAPT composed of acetylsalicylic acid + clopidogrel up to 6M. Then, continue with acetylsalicylic acid.
  Interventions: Device: Xience: Everolimus-eluting stent; Drug: 12-month DAPT (Standard of care)

INTERVENTIONS:
Device: Angiolite: Sirolimus-eluting stent — The angiolite stent (iVascular, Barcelona, Spain) is a thin-strut cobalt-chromium sirolimus-eluting stent with an open-cell design containing a durable biostable coating composed of three layers - acrylate to ensure adhesion to the metal surface, fluoroacrylate that carries the sirolimus, and a top layer of fluoroacrylate to control drug release.
  Other Names: iVascular angiolite
  Arms: Angiolite and abbreviated DAPT; Angiolite and standard of care DAPT
Device: Xience: Everolimus-eluting stent — The Xience stent family (Abbott vascular, California, United States of America), characterized by an L-605 cobalt-chromium (CoCr) is a thin-strut cobalt-chromium everolimus-eluting stent with an open-cell design containing a nonerodable polymer made of PBMA, a reservoir made of a fluorinated copolymer of vinylidene fluoride and hexafluoropropylene monomers. Xience™ stent family includes XIENCE Skypoint™ and XIENCE Sierra™
  Other Names: Xience stent family
  Arms: Xience stent family and abbreviated DAPT; Xience stent family and standard of care DAPT
Drug: 1-month DAPT — DAPT with acetylsalicylic acid + prasugrel or ticagrelor for 1 month. Then, only the same oral P2Y12 inhibitor (clopidogrel, prasugrel, and ticagrelor) up to 12 months.
  The type of agent and treatment duration will be selected according to the clinical characteristic of the patient: Acute coronary syndrome or Chronic coronary syndrome and Need for OAC or No need for OAC
  Arms: Angiolite and abbreviated DAPT; Xience stent family and abbreviated DAPT
Drug: 12-month DAPT (Standard of care) — DAPT with acetylsalicylic acid and prasugrel or ticagrelor up to 12 months. The type of agent and treatment duration will be selected according to the clinical characteristic of the patient: Acute coronary syndrome or Chronic coronary syndrome and Need for OAC or No need for OAC
  Arms: Angiolite and standard of care DAPT; Xience stent family and standard of care DAPT

SUMMARY:
Factorial 2x2, all-comer, multicentre, randomized controlled trial (ratio 1:1:1:1). First, the study will compare (first randomization) the non-inferiority in target lesion failure of angiolite stent versus Xience stent family. Immediately after the first randomization, the study compares (second randomization) the superiority in bleeding Bleeding Academic Research Consortium (BARC) 2, 3, or 5 of abbreviated DAPT versus standard of care. Both primary endpoints will be evaluated at 12 months of follow-up. The study will be open-label for the stent type and the antiplatelet regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 - < 95 years;
* Presence of one or more coronary artery stenosis of 50% or more in a native coronary artery or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation. The vessel should have a reference vessel diameter of at least 2.00 mm (no limitation on the number of treated lesions, vessels, or lesion length);
* Able to provide informed consent and willing to participate in the trial.

Exclusion Criteria:

* Known intolerance to acetylsalicylic acid, P2Y12 inhibitors (clopidogrel, prasugrel, or ticagrelor), sirolimus, everolimus, or chromium-cobalt.;
* Known severe hepatic impairment Child-Pug stage C;
* Prior PCI (not related to the study) performed in the last 45 days;
* Planned non-cardiac surgery during the first month after PCI, unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
* Planned coronary artery bypass graft (CABG) or any other cardiac surgery (valvular for instance) following index PCI;
* Active major bleeding or major surgery within the last 30 days;
* Known stroke (any type) within the 30 days prior to the randomization;
* Women of childbearing potential being defined as woman from the onset of menstruation (menarche) until they become postmenopausal, unless they are permanently sterile. A postmenopausal state is clarified as having no menstrual periods for 12 consecutive months without any other medical cause. Women who have undergone permanent sterilization methods, including hysterectomy, bilateral salpingectomy, and bilateral oophorectomy, can be enrolled in the study
* Currently participating in another randomized controlled trial and not yet at its primary endpoint;
* Life expectancy less than one year due to non-cardiovascular comorbidity.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2312 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
To determine the rate of target lesion failure between angiolite stent and Xience stent family (tested for non-inferiority) in both the standard of care DAPT regimen and abbreviated antiplatelet therapy group. | 1 year
To determine the rate of clinically relevant bleeding events (BARC 2, 3, or 5) between an abbreviated DAPT regimen and the standard of care DAPT (tested for superiority of the experimental arm). | 1 year

SECONDARY OUTCOMES:
To determine the rate of adverse ischemic events between an abbreviated dual antiplatelet therapy regimen and the standard of care dual antiplatelet therapy (tested for non-inferiority). | 1 year
Rate of target lesion failure between angiolite stent and Xience stent family (Skypoint or Sierra) (tested for non-inferiority) in the standard of care subgroup. | 1 year

OTHER OUTCOMES:
To determine the rate of Patient-Oriented Composite endpoint | 1-2-3-4-5 years
To determine the rate of individual components of All cause, cardiovascular, and cardiac death | 1-2-3-4-5 years
To determine the rate of recurrent myocardial infarction | 1-2-3-4-5 years
To determine the rate of target lesion revascularization | 1-2-3-4-5 years
To determine the rate of target vessel revascularization | 1-2-3-4-5 years
To determine the rate of stent thrombosis | 1-2-3-4-5 years
To determine the rate of clinical device success | Immediatly after the procedure
To determine the rate of clinical procedural success | Immediatly after the procedure
To determine the rate of bleeding events | 1-2-3-4-5 years
To determine the rate of net adverse clinical endpoints (NACE) | 1-2-3-4-5 years
To determine the rate of major adverse cardiac and cerebral events (MACCE) | 1-2-3-4-5 years
To determine the rate of transfusion rates | 1-2-3-4-5 years
To determine the rate of clinically relevant bleeding events (BARC 2, 3, or 5) at 1 year between an abbreviated dual antiplatelet therapy regimen and the standard of care dual antiplatelet therapy in the female population of the study | 1 year
To determine the rate of adverse ischemic events at 1 year between an abbreviated dual antiplatelet therapy regimen and the standard of care dual antiplatelet therapy in the female population of the study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabaté, Principal Investigator — Hospital Clinic of Barcelona
Locations (39):
- Belgium (9):
  - Olv Aalst, Aalst
  - IMELDA, Bonheiden
  - CHU Marie Curie, Charleroi
  - ZOL GENK, Genk
  - CHC Montlégia, Liège
  - Hospital de La Citadelle, Liège
  - Chu Ambroise Pare, Mons
  - Az Delta, Roeselare
  - Az Turnhout, Turnhout
- France (4):
  - Chu Lille, Lille
  - Icps Massy, Massy
  - Ipcs Quincy, Quincy-sous-Sénart
  - Chu Toulouse, Toulouse
- Spain (26):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Vall D'Hebrón, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Jerez de La Frontera, Jerez de la Frontera
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Clínico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza